CLINICAL TRIAL: NCT00183820
Title: A Phase II Study of Gemcitabine, Oxaliplatin, and Paclitaxel in Patients With Refractory Germ Cell Carcinoma
Brief Title: Study of Gemcitabine, Oxaliplatin, and Paclitaxel in Patients With Refractory Germ Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4T-03-1
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Testicular Cancer; Germ Cell Neoplasm
Keywords: Testicular; Extra gonadal germ cell neoplasm
MeSH Terms: conditions — Testicular Neoplasms; Neoplasms, Germ Cell and Embryonal | interventions — Paclitaxel; Gemcitabine; Oxaliplatin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: paclitaxel, gemcitabine, and oxaliplatin

INTERVENTIONS:
Drug: paclitaxel, gemcitabine, and oxaliplatin — 1. Paclitaxel 170 mg/m2 IV d 1 14 days
  2. Gemcitabine 800 mg/m2 IV d 1 14 days
  3. Oxaliplatin 100 mg/m2 IV d 1 14 days

SUMMARY:
This is a study for patients with advanced testicular cancer. This research study involves treatment with oxaliplatin, paclitaxel, and gemcitabine, which is an investigational chemotherapy combination. This study is for patients who have not responded to standard cisplatin-containing chemotherapy or the cancer has returned after such treatment.

This research is being done to assess the effectiveness of the proposed combination of medications for this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Prior histologic or serologic confirmation of testicular or extragonadal germ cell neoplasm not amenable to surgical cure
2. Must have refractory germ cell neoplasm defined as one or more of the following:

   * patients who progress during or within 4 weeks of cisplatin-containing tx, OR - patients who have failed initial salvage chemotx regimens, including high-dose tx (chemotx with stem cell support), POMB-ACE tx, VeIP, or VIP
3. Must have one or more of the following (check all that apply):

   * unidimensionally measurable doze assessed within 14 days prior to registration,
   * elevated β-HCG > 20 mIU assessed within 24-48 hours prior to registration, OR
   * AFP > 2 x uln assessed within 5-7 days prior to registration

   Note: Soft tissue dz, which has been radiated in the 2 months prior to registration, is not assessable as measurable dz.
4. X-rays, scans, or PE for non-measurable dz must have been completed within 14 days of registration
5. May have received prior surgery or RT. At least 3 weeks must have elapsed since completion of previous tx and must have recovered from any adverse effects
6. Zubrod PS less than or equal to 2
7. Greater than or equal to 16 years of age
8. AGC greater than or equal to 1.5; platelets greater than or equal to 100,000
9. Total bilirubin < 2.5 x uln; SGOT and alk phos < 5 x uln (obtained within 14 days prior to registration)
10. LDH (obtained within 7 days prior to registration)
11. Creatinine < 2.5 x uln or calc or meas CrCl greater than or equal to 40 ml/min (obtained within 14 days prior to registration; patient must not be on renal dialysis)
12. Serum K+ and Mg++ within inst range of normal (obtained within 14 days prior to registration)
13. Men of reproductive potential must agree to use effective contraceptive method
14. Signed informed consent (including HIPAA authorization)

Exclusion Criteria:

1. Prior tx with cytotoxic or experimental agents within 14 days prior to registration
2. Evidence of concurrent infection (T > 96.8F but < 101.5F; WBC < 11.0 unless these values can be ascribed to another tumor-related phenomena)
3. Other prior malignancy, except adequately treated basal cell or squamous cell skin cancer, adequately treated stage I or II cancer from which patient is currently in chemoradiation (CR), or any other cancer from which patient has been disease-free for 5 years

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-11; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Tumor Response | Every 6 weeks

SECONDARY OUTCOMES:
Progression | Every 9 wks

CONTACTS AND LOCATIONS:
Overall Officials: David Quinn, MD, Principal Investigator — University of Southern California
Locations (1):
- Norris Comprehensive Cancer Center, Los Angeles, California, United States